CLINICAL TRIAL: NCT07341737
Title: A Phase 1/2, Multicentre, Open-Label, Dose Escalation and Expansion Study to Assess the Safety, Pharmacokinetics, and Preliminary Efficacy of SL-28 in Patients With Advanced Solid Tumours
Brief Title: SL-28 for Advanced Solid Tumours
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Second Life Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SL-28-FIH
Record Dates: First submitted 2025-11-17; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Head & Neck Cancer; Pancreas Carcinoma; Pancreas Cancer, Metastatic; Lung Adenocarcinoma; Lung Cancer (NSCLC); Lung Cancer (Non-Small Cell); Esophageal Cancer; Stomach (Gastric) Cancer; Liver Cancer; Intestinal Cancer; Bladder Cancer; Renal Cancer; Prostate Cancer; Melanoma (Skin Cancer); Breast Cancer; Ovarian Cancer; Endometrial Cancer; Colorectal Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Pancreatic Neoplasms; Neoplasm Metastasis; Adenocarcinoma of Lung; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Stomach Neoplasms; Liver Neoplasms; Intestinal Neoplasms; Urinary Bladder Neoplasms; Kidney Neoplasms; Prostatic Neoplasms; Melanoma; Breast Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a Phase 1/2 open-label study to assess the safety, pharmacokinetics (PK), and preliminary efficacy of SL-28, an allogeneic, non human leukocyte antigen (HLA)-matched, modified T -cell-based treatment for advanced and unresectable solid tumours.
  The study will be conducted in 4 parts:
  * Part 1: Phase 1a dose escalation as a 3+3 design, with a single dose on Day 1 followed by daily dosing from Day 8
  * Part 2: Phase 1b dose expansion at the maximum tolerated dose (MTD)
  * Part 3: Phase 2a dose expansion in 3 tumour types
  * Part 4: Phase 2a dose expansion in the tumour type showing the highest efficacy to SL-28
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SL-28 Low Dose (Experimental)
  Interventions: Biological: SL-28
- SL-28 Intermediate Dose (Experimental)
  Interventions: Biological: SL-28
- SL-28 High Dose (Experimental)
  Interventions: Biological: SL-28

INTERVENTIONS:
Biological: SL-28 — Doses administered: 3×10^7 cells/injection, once daily, 5 days per week, 12 weeks.
  Mode of administration: intravenous push
  Arms: SL-28 Low Dose
Biological: SL-28 — Doses administered: 6×10^7 cells/injection, once daily, 5 days per week, 12 weeks.
  Mode of administration: intravenous push
  Arms: SL-28 Intermediate Dose
Biological: SL-28 — Doses administered: to-be-determeined-later Mode of administration: intravenous push
  Arms: SL-28 High Dose

SUMMARY:
Second Life Therapeutics is developing SL-28, an allogeneic, non-genetically modified cell-based therapy for the treatment of advanced solid tumours. The company has recently demonstrated a novel, non-genetic approach to modulate immune cell activity through targeted manipulation of the Universal Receptive System. The purpose of this open label, multi-center clinical trial is to evaluate the anti-tumor activity, safety, and pharmacokinetics, single-agent SL-28 in patients with a diverse array of solid tumors. The study includes an initial Phase 1 dose escalation to determine recommended dose(s) for expansion of SL-28 as a monotherapy and Phase 2 expansion cohorts. The study will enroll patients with advanced solid tumours, including those who failed previous lines of chemo- and immunotherapies.

DETAILED DESCRIPTION:
This study aims to assess the anti-tumour activity, safety, and interactions of single-agent SL-28 as an anti-cancer treatment in patients with a diverse array of solid tumours.

Who is it for? You may be eligible for this study if you are aged 18 years or older, you have been diagnosed with advanced solid tumor, including head and neck cancer, small-cell lung cancer, non-small cell lung cancer; mesothelioma; oesophageal cancer, gastric cancer, liver cancer, colorectal cancer, pancreatic cancer, bladder cancer, kidney cancer, prostate cancer, ovarian cancer, endometrial cancer, breast cancer or skin cancer (melanoma) that is locally advanced, metastatic or unable to be surgically removed. Patients will also be assessed by a study doctor to ensure that they are well enough to participate in the trial before they will be offered enrolment into the study.

Study details All participants who choose to enroll in this study will receive 12 weeks of SL-28 treatment, administered on a 5-days-on, 2-days-off schedule. The first group of participants to receive SL-28 will be monitored for 12 weeks before a second group may be administered a higher dose of SL-28. Up to three cohorts will be enrolled to determine the highest safe and effective dose that does not cause severe side effects in patients.

It is hoped this study will show that SL-28 is safe to deliver to patients with solid tumour cancers, and determine the highest dose of SL-28 that cancer patients can safely receive.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent prior to any study-related procedures and to understand the nature, purpose, and potential risks of the study
* Adult males and females ≥18 years of age at screening
* Life expectancy of at least 3 months
* Histologically or cytologically confirmed unresectable advanced solid tumor (recurrent, metastatic, or locally advanced)
* Disease refractory to, intolerant of, or refusal of standard therapies, including immunotherapy and molecular/biomarker-directed treatments, as determined by the Principal Investigator (PI) or delegate
* Eligible tumor types include:
* Head and neck squamous cell carcinoma
* Thoracic malignancies (small-cell lung cancer, non-small cell lung cancer, esophageal cancer)
* Gastrointestinal malignancies (gastric, liver, colorectal, pancreatic adenocarcinoma)
* Genitourinary malignancies (bladder, renal cell, prostate cancer)
* Gynecologic malignancies (ovarian, endometrial cancer)
* Breast cancer and melanoma
* Evaluable disease per RECIST v1.1
* ECOG performance status 0-1 (or up to 2 at PI discretion)
* Adequate organ function, defined as:
* Total bilirubin ≤1.5 × ULN (≤2.0 × ULN for liver metastases or Gilbert's syndrome)
* AST, ALT, alkaline phosphatase ≤2.5 × ULN (≤5 × ULN if liver metastases, at PI discretion)
* Creatinine clearance ≥50 mL/min (Cockcroft-Gault) or eGFR ≥50 mL/min (CKD-EPI)
* Absolute neutrophil count ≥1,000/mm³
* Platelet count ≥100,000/mm³
* Hemoglobin ≥90 g/L without transfusion within 2 weeks
* Prothrombin time and aPTT ≤1.5 × ULN (or stable INR if on anticoagulation)

Female patients:

-Non-childbearing potential (surgically sterile or postmenopausal), or of childbearing potential with negative pregnancy tests and agreement to effective contraception through 90 days post-dose

Male patients:

* Agreement not to donate sperm for 90 days post-dose
* Agreement to use adequate contraception as applicable
* Suitable venous access for blood sampling
* Willingness and ability to comply with study procedures and protocol requirements

Exclusion Criteria:

* Ongoing toxicities ≥ Grade 2 per NCI CTCAE v5.0 (except alopecia, fatigue, sensory neuropathy, or adequately treated endocrine deficiencies)
* NYHA Class III or IV heart disease, myocardial infarction within 6 months, unstable arrhythmia, or ischemia on ECG
* QTcF >470 ms (females) or >450 ms (males)
* Active, uncontrolled bacterial, viral, or fungal infection requiring systemic therapy
* Requirement for systemic corticosteroids or other immunosuppressive therapy that cannot be discontinued ≥14 days prior to dosing
* Prior therapies within restricted timeframes:
* Immune checkpoint inhibitors or biologics within 28 days
* Antineoplastic therapies, surgery, radiotherapy, or radiopharmaceuticals within 21 days
* Unapproved investigational drugs within 5 half-lives
* Nitrosoureas or mitomycin C within 6 weeks
* Concurrent malignancy within 5 years, except specified low-risk cancers
* Pregnancy or breastfeeding
* Known HIV, hepatitis B (HBsAg positive), or hepatitis C infection
* Inability or unwillingness to comply with protocol procedures
* History of anaphylaxis or significant allergy interfering with participation
* Clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, neurologic, psychiatric, or immunologic disease within 6 months
* Conditions affecting drug absorption, distribution, metabolism, or excretion
* Receipt of live vaccines within 28 days prior to screening
* Participation in another investigational study within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events | 12 weeks
  Treatment-emergent adverse events will be assessed and graded by the investigator according to the CTCAE v5
To evaluate the safety and tolerability of SL-28 by determining the incidence of dose-limiting toxicitieswithin the first 28 days after infusion. | 12 weeks
  Assessment of dose limiting toxicities assessed by the occurrence of treatment-emergent adverse events(TEAEs) graded by the Investigator per the National Cancer Institute Common Terminology Criteria forAdverse Events, version 5.0.
Change from baseline in ECG QT interval | 12 weeks
  Electrocardiograms will be recorded using a 12-lead ECG machine, and the QT interval (milliseconds) will be evaluated and summarized as change from baseline.
Change from baseline in vital signs | 12 weeks
  Vital signs including systolic blood pressure (mmHg) and diastolic blood pressure (mmHg)will be measured using standard clinical equipment and summarized as change from baseline.
Change from baseline in vital signs | 12 weeks
  Vital signs: Heart rate (beats per minute) will be measured using standard clinical equipment and summarized as change from baseline.
Change from baseline in vital signs | 12 weeks
  Vital signs: body temperature (°C) will be measured using standard clinical equipment and summarized as change from baseline.
Number of participants with dose-limiting toxicities (DLTs) | 12 weeks
  Dose-limiting toxicities will be assessed during the DLT evaluation period as defined in the protocol.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per RECIST 1.1 | 12 weeks
  Objective response rate will be defined as the proportion of participants achieving a complete response (CR) or partial response (PR) according to RECIST version 1.1, as assessed by CT or MRI imaging.
Objective Response Rate (ORR) per iRECIST | 12 weeks
  Objective Response Rate (ORR) per iRECIST
Disease Control Rate (DCR) per RECIST 1.1 | 12 weeks
  Disease control rate will be defined as the proportion of participants achieving CR, PR, or stable disease (SD) according to RECIST version 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Hollywood Private Hospital, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tetz V, Kardava K, Shulenbayev O, Vecherkovskaya M, Khodadadi-Jamayran A, Tsirigos A, Tetz G. Partial response in a patient with skeletal and hepatic metastases following resected pancreatic cancer to the novel cell therapy SL-28: a case report. Front Oncol. 2025 Nov 19;15:1636989. doi: 10.3389/fonc.2025.1636989. eCollection 2025. PMID 41347084
- [Background] Tetz V, Kardava K, Shulenbayev O, Vecherkovskaya M, Khodadadi-Jamayran A, Tsirigos A, Tetz G. Dramatic Clinical Response to a Novel Form of Cell Therapy SL-28 in a Patient with Prostate Cancer and Bone Metastasis: A Case Report. Immunotargets Ther. 2025 Oct 29;14:1201-1207. doi: 10.2147/ITT.S547989. eCollection 2025. PMID 41185720
- [Background] Tetz V, Tetz G. Novel prokaryotic system employing previously unknown nucleic acids-based receptors. Microb Cell Fact. 2022 Oct 4;21(1):202. doi: 10.1186/s12934-022-01923-0. PMID 36195904
- [Background] Tetz V, Kardava K, Vecherkovskaya M, Khodadadi-Jamayran A, Tsirigos A, Tetz G. Regulating white blood cell activity through the novel Universal Receptive System. bioRxiv [Preprint]. 2025 Jan 20:2025.01.06.631232. doi: 10.1101/2025.01.06.631232. PMID 39896476
- [Background] Tetz G, Kardava K, Vecherkovskaya M, Khodadadi-Jamayran A, Tsirigos A, Tetz V. Universal receptive system as a novel regulator of transcriptomic activity of Staphylococcus aureus. Microb Cell Fact. 2025 Jan 3;24(1):1. doi: 10.1186/s12934-024-02637-1. PMID 39754239
- [Background] Tetz V, Kardava K, Vecherkovskaya M, Khodadadi-Jamayran A, Tsirigos A, Tetz G. The universal receptive system: a novel regulator of antimicrobial and anticancer compound production by white blood cells. J Leukoc Biol. 2025 Jun 4;117(6):qiaf085. doi: 10.1093/jleuko/qiaf085. PMID 40578310